CLINICAL TRIAL: NCT07244835
Title: A First in Human Phase 1 Open-Label, Multicenter, Dose Escalation and Expansion Study of DEG6498 in Patients With Solid Tumors
Brief Title: A Study of DEG6498 in Participants With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Degron Therapeutics Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DEG6498-ONC-2401
Record Dates: First submitted 2025-11-13; First posted 2025-11-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Malignant Neoplasms
Keywords: DEG6498; Solid tumor; Phase 1; BRAF mutation; Hepatocellular carcinoma (HCC); Melanoma; Colorectal cancer (CRC); Lung cancer; Thyroid cancer; Ovarian cancer; Pancreatic cancer; Glioblastoma; Renal cancer; Malignant peripheral nerve sheath tumor (MPNST)
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular; Melanoma; Colorectal Neoplasms; Lung Neoplasms; Thyroid Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Glioblastoma; Kidney Neoplasms; Neurofibrosarcoma

STUDY DESIGN:
Intervention Model Description: This is a dose escalation and dose expansion Ph1 study. In dose escalation part, participants in single arms will receive DEG6498 capsules daily from a starting dose with dose escalation decision made at a 3+3 model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DEG6498 Treatment (Experimental): Participants in dose escalation part will receive DEG6498 capsules orally once a day in each treatment cycle of 28 days at different ascending dose level.
  Participants in dose expansion part will receive DEG6498 capsules orally once a day in each treatment cycle of 28 days at a dose level decided based on dose escalation results.
  Interventions: Drug: DEG6498

INTERVENTIONS:
Drug: DEG6498 — DEG6498 is an orally bioavailable molecular glue drug that potently induces the degradation of human antigen R (HuR).

SUMMARY:
The goal of this first in human, Phase 1, multi-center, open-label, and 2-part study is to learn whether DEG6498 is safe and tolerable in participants with advanced solid tumors. It will also learn about DEG6498 pharmacokinetics (PK) profile and potential antitumor activity. The main questions it aims to answer are:

* what is an appropriate dose to be given to participants?
* are the side effects of treatment manageable?

Participants who are treated in this study will receive DEG6498 orally once a day and be closely monitored by the treating physicians.

DETAILED DESCRIPTION:
This study will be conducted in 2 Parts. Part 1, the dose escalation part of the study, will test different doses of DEG6498 as a single agent when administered to participants with any type of advanced solid tumor that has no available alternative treatments, and determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) for further studies. Part 2, the dose expansion part of the study, will further characterize the safety/tolerability profile and clinical activities of DEG6498 in 2 tumor types: BRAF mutant tumors and hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for the study prior to the performance of any study-specific procedures
2. Male and female older than or equal to 18 years of age at the time signing the informed consent form (ICF)
3. If female, must be postmenopausal, or surgically sterile, or agree to highly effective contraceptive measures to prevent pregnancy throughout treatment period and within 30 days of last study drug treatment
4. Women of childbearing potential (WOCBP) must have 2 negative pregnancy tests (1 serum test required) as verified by the investigator prior to starting study drug
5. If male, must agree to inform and ensure their female partners to use highly effective contraception measures to prevent pregnancy, and to refrain from donating sperm while on study drug and for at least 30 days following DEG6498 discontinuation
6. Patients with advanced solid tumors, who have failed standard therapies, or for whom no standard therapy exists

   1. Part 1: Advanced solid tumor patients
   2. Part 2: Patients with BRAF mutation positive tumors and HCC
7. Presence of at least 1 measurable lesion according to RECIST v1.1 .
8. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

1. Participant has a significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study, puts the participant at unacceptable risk if he/she were to participate in the study
2. Participant has a condition that confounds the ability for interpret data from the study
3. Pregnant or breastfeeding women
4. Active or concurrent malignancy requiring treatment (including both systemic therapy and radiotherapy) within 14 days or 5 half lives (whichever is shorter) prior to the first dose of study drug, or received antibody therapy within 28 days
5. Symptomatic CNS metastases which are neurologically unstable, or CNS metastases requiring local CNS directed therapy, or increasing doses of corticosteroids within 2 weeks of first dose of study treatment.
6. Clinically significant cardiovascular disease
7. Known active or chronic infection that requires systemic therapy within 2 weeks of first dose of study drug
8. Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome, or active HBV or HCV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | From first dose through the end of Cycle 1 (each cycle is 28 days)
  Number of participants with DLT in Part 1
Incidence of adverse events (AEs) and serious AEs (SAEs) as assessed by CTCAE v5.0 | From Screening up to 30 days after the last dose
  Number, type, frequency, severity, timing, and relationship to DEG6498 of AEs, SAEs, etc

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) of DEG6498 | From Day 1 in Cycle 1 followed by Day 1 of each treatment cycle through treatment until EOT visit, expected average 6 months (each cycle is 28 days)
  Measurement of plasma concentration over time for exposure to DEG6498
Maximum concentration (Cmax) of DEG6498 | From Day 1 in Cycle 1 followed by Day 1 of each treatment cycle through treatment until EOT visit, expected average 6 months (each cycle is 28 days)
  Measurement of plasma concentration over time for exposure to DEG6498
Time to reach maximum concentration (Tmax), | From Day 1 in Cycle 1 followed by Day 1 of each treatment cycle through treatment until EOT visit, expected average 6 months (each cycle is 28 days)
  Measurement of plasma concentration over time for DEG6498 to reach maximum concentration
Terminal half-life (T1/2) of DEG6498 | From Day 1 in Cycle 1 followed by Day 1 of each treatment cycle through treatment until EOT visit, expected average 6 months (each cycle is 28 days)
  Measurement of the clearance of DEG6498 from plasma over time
Clearance following oral dose (CL/F) of DEG6498 | From Day 1 in Cycle 1 followed by Day 1 of each treatment cycle through treatment until EOT visit, expected average 6 months (each cycle is 28 days)
  Measurement of the clearance of DEG6498 from plasma over time
Overall response rate (ORR) | From the date of dosing until the date of first documented progression, unacceptable toxicity, death from any cause, participant withdraw consent, or investigator's decision, whichever occurs first, expected up to 30 months
  The proportion of participants with best overall response of complete response (CR) or partial response (PR) as determined by the Investigator per RECIST 1.1
Time to response (TTR) | From the date of dosing until the date of first documented progression, unacceptable toxicity, death from any cause, participant withdraw consent, or investigator's decision, whichever occurs first, expected up to 30 months
  The time interval from the first DEG6498 dose date to the date of first documented objective response
Disease control rate (DCR) | From the date of dosing until the date of first documented progression, unacceptable toxicity, death from any cause, participant withdraw consent, or investigator's decision, whichever occurs first, expected up to 30 months
  The proportion of participants with a best ORR + Stable Disease (SD)
Duration of response (DOR) | From the date of dosing until the date of first documented progression, unacceptable toxicity, death from any cause, participant withdraw consent, or investigator's decision, whichever occurs first, expected up to 30 months
  The time interval from the earliest occurrence of a documented objective response to the first time of disease progression or death from any cause, whichever comes first

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No